CLINICAL TRIAL: NCT00896051
Title: TMC125-TiDP2-C238: A Randomized, Exploratory, Open-label 48-week Trial to Investigate the Pharmacokinetics, Safety, Tolerability and Antiviral Activity of Etravirine (ETR) in Combination With Ritonavir-boosted Atazanavir (ATV/Rtv) and 1 NRTI in Treatment-experienced HIV-1 Infected Subjects
Brief Title: TMC125-TiDP2-C238: An Exploratory Pharmacokinetics, Safety and Anti-HIV Activity Study of Etravirine (ETR) When Given With Boosted Atazanavir (ATV/Rtv) at Two Different Doses and 1 Nucleoside Reverse Transcriptase Inhibitor (NRTI) in Treatment Experienced HIV Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016045; TMC125-TiDP2-C238 (Other: Janssen R&D Ireland)
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: HIV Infections; Acquired Immunodeficiency Syndrome; TMC125-TiDP2-C238; TMC125-C238; Etravirine; Intelence; HIV; HIV-1; Pharmacokinetics
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Atazanavir Sulfate; Ritonavir; Reverse Transcriptase Inhibitors; etravirine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATV/rtv 300/100 mg (Treatment A) (Experimental): Treatment-experienced human immunodeficiency virus - type 1 (HIV-1) infected participants will take by mouth atazanavir (ATV)/low-dose ritonavir (rtv) 300/100 mg once daily + 2 nucleoside reverse transcriptase inhibitors (NRTIs) for 2 weeks pre-treatment followed by ATV/rtv 300/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 NRTI for 48 weeks. If particpating in an optional substudy to assess the effect of adding tenofovir disoproxil fumarate (TDF) for 7 days on ATV and ETR pharmacokinetics, participants will receive TDF 300 mg once daily for 7 days in addition to their antiretroviral regimen (ETR+ATV/rtv+NRTI).
  Interventions: Drug: Atazanavir (ATV) 300 mg; Drug: Ritonavir (rtv) 100 mg; Drug: Nucleo(side)/(tide) reverse transcriptase inhibitors (NRTIs); Drug: Etravirine (ETR) 200 mg; Drug: Tenofovir disoproxil fumarate (TDF) 300 mg
- ATV/rtv 400/100 mg (Treatment B) (Experimental): Treatment-experienced human immunodeficiency virus - type 1 (HIV-1) infected participants will take by mouth atazanavir (ATV)/low-dose ritonavir (rtv) 300/100 mg once daily + 2 nucleoside reverse transcriptase inhibitors (NRTIs) for 2 weeks pretreatment followed by ATV/rtv 400/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 NRTI for 48 weeks. If particpating in an optional substudy to assess the effect of adding tenofovir disoproxil fumarate (TDF) for 7 days on ATV and ETR pharmacokinetics, participants will take TDF 300 mg once daily for 7 days in addition to their antiretroviral regimen (ETR+ATV/rtv+NRTI).
  Interventions: Drug: Atazanavir (ATV) 400 mg; Drug: Ritonavir (rtv) 100 mg; Drug: Nucleo(side)/(tide) reverse transcriptase inhibitors (NRTIs); Drug: Etravirine (ETR) 200 mg; Drug: Tenofovir disoproxil fumarate (TDF) 300 mg

INTERVENTIONS:
Drug: Atazanavir (ATV) 300 mg — Atazanavir (ATV) 300 mg taken by mouth following a meal each morning for 2 weeks during the Pre-Treatment Period and for 48 weeks during the Treatment Period. If participating in the optional substudy, participants will take ATV 300 mg by mouth following a meal each morning on Substudy Days -1 to 7.
  Arms: ATV/rtv 300/100 mg (Treatment A)
Drug: Atazanavir (ATV) 400 mg — Atazanavir (ATV) 400 mg taken by mouth following a meal each morning for 2 weeks during the Pre-Treatment Period and for 48 weeks during the Treatment Period. If participating in the optional substudy, participants will take ATV 400 mg by mouth following a meal each morning on Substudy Days -1 to 7.
  Arms: ATV/rtv 400/100 mg (Treatment B)
Drug: Ritonavir (rtv) 100 mg — Ritonavir (rtv) 100 mg taken by mouth following a meal each morning for 2 weeks during the Pre-Treatment Period and for 48 weeks during the Treatment Period. If participating in the optional substudy, participants will take rtv 100 mg by mouth following a meal each morning on Substudy Days -1 to 7.
Drug: Nucleo(side)/(tide) reverse transcriptase inhibitors (NRTIs) — 2 investigator-selected NRTIs taken as specified in the individual product labels for 2 weeks during the Pre-Treatment Period followed by 1 investigator-selected NRTI (of the 2 NRTIs in the Pre-Treatment Phase) taken as specified in the individual product label for 48 weeks during the Treatment Period. If participating in the optional substudy, participants will take 1 investigator-selected NRTI (of the 2 NRTIs in the Pre-Treatment Phase) mg taken as specified in the individual product label during the Substudy.
Drug: Etravirine (ETR) 200 mg — Etravirine (ETR) 200 mg taken twice daily as two 100-mg tablets following a meal (morning and evening) for at least the first two weeks of the 48-week Treatment Period. If participating in the optional substudy, participants will take ETR 200 mg twice daily as two 100-mg tablets following a meal each morning and evening on Substudy Days -1 to 7.
Drug: Tenofovir disoproxil fumarate (TDF) 300 mg — Tenofovir disoproxil fumarate (TDF) 300 mg taken by mouth following a meal each morning on Substudy Days 1 to 7.

SUMMARY:
The purpose of this study is to determine the pharmacokinetics (how the body absorbs, distributes, metabolizes and eliminates a drug) (PK) of ETR when given with ATV/rtv and 1 NRTI in treatment experienced HIV-1 infected patients. In addition, safety, tolerability and anti-HIV effect of this regimen will also be studied. A total of 46 patients will be enrolled.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), exploratory, open-label (all involved people know the identity of the intervention) trial to evaluate the pharmacokinetics (PK), safety, tolerability and anti-HIV (anti Human Immunodeficiency Virus) activity of etravirine (ETR ) when given with atazanavir/ritonavir (ATV/rtv) and 1 nucleoside reverse transcriptase inhibitor (NRTI) in 46 treatment experienced HIV-1 infected patients. The trial will consist of : 4 weeks of Screening Period, 2 weeks Pre-Treatment Phase, 48-week Treatment Period, and a Final Visit followed by a 4-week Follow-up Period (only for patients not continuing treatment with ETR in another trial or program). Safety evaluations (AE reporting, labs, vital signs, etc.) will be monitored at each study visit. A PK substudy (included in the protocol, with optional participation) with tenofovir (TDF) added to the antiretroviral regimen for 7 days will be conducted in patients with > 24 weeks of treatment with suppressed HIV-1 viral load. In Pre-Treatment Phase, all patients will receive ATV/rtv 300/100 mg once daily to be taken following a meal each morning + 2 NRTIs (dose as specified in the labels) for 14 days. In Treatment Phase, patients will receive ETR 200 mg twice daily in addition to ATV/rtv (300/100 mg or 400/100 mg) once daily with meals + 1 investigator-selected NRTI for 48 weeks. In substudy TDF 300 mg once daily will be added to the treatment regimen x 7 days.

ELIGIBILITY:
Inclusion Criteria:

- Documented HIV-1 infection

* Failing on a stable ART (anti retroviral therapy) with HIV-1 plasma viral load above 500 HIV-1 RNA copies/ml
* Presence of at least 1 documented NNRTI mutation
* Demonstrated sensitivity to ATV, ETR and at least one of the selected NRTIs based on the resistance test at screening
* General medical condition, in the investigator's opinion, does not interfere with the assessments and completion of the trial
* Substudy: patients who have been treated in C238 for more than 24 weeks and are currently suppressed (defined as patients with at least 2 most recent and consecutive viral loads less than 50 cp/mL) will be considered eligible for the substudy

Exclusion Criteria:

* Primary HIV-1 infection
* Previously documented HIV-2 infection
* Previously failed 2 or more HIV PI-containing regimens
* Previous diagnosis of hereditary hyperbilirubinemia (eg. Gilbert's syndrome, Crigler-Najjar syndrome).

Grade 3 or 4 toxicities (according to DAIDS grading)

* Acute and chronic viral hepatitis
* Receipt of an investigational drug or investigational vaccine within 30 days prior to the trial drug administration
* Pregnant or breastfeeding female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (18):
- United States (10):
  - Little Rock, Arkansas
  - Bakersfield, California
  - Beverly Hills, California
  - Orlando, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Macon, Georgia
  - Dallas, Texas
  - Houston, Texas
- Argentina (2):
  - Buenos Aires
  - Córdoba
- France (2):
  - Paris
  - Tourcoing
- South Africa (3):
  - Bloemfontein
  - Cape Town
  - George
- Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Etravirine coadministered with 2 doses of atazanavir/low-dose ritonavir each combined with 1 nucleoside reverse transcriptase inhibitor was evaluated in human immunodeficiency virus - type 1 infected participants. The study was conducted between 25 June 2009 and 10 April 2012 and participants were recruited by 17 investigators in 4 countries.
Pre-assignment Details: Fifty (50) participants were enrolled in the study and received treatment with study drug during a 2-week Pre-treatment Period (Week -2 to Day -1) and a 48-week Treatment Period (Day 1 to Week 48). Efficacy data are reported for the 48-week Treatment Period.
Groups:
- ATV/Rtv 300/100 mg (Treatment A): Treatment-experienced human immunodeficiency virus - type 1 (HIV-1) infected participants took by mouth atazanavir (ATV)/low-dose ritonavir (rtv) 300/100 mg once daily + 2 nucleoside reverse transcriptase inhibitors (NRTIs) for pre-treatment for 2 weeks followed by ATV/rtv 300/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 NRTI for 48 weeks.
- ATV/Rtv 400/100 mg (Treatment B): Treatment-experienced human immunodeficiency virus - type 1 (HIV-1) infected participants took by mouth atazanavir (ATV)/low-dose ritonavir (rtv) 300/100 mg once daily + 2 nucleoside reverse transcriptase inhibitors (NRTIs) pretreatment for 2 weeks followed by ATV/rtv 400/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 NRTI for 48 weeks.
Period: Overall Study
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment B)
Started | 25 | 25
Completed | 15 | 16
Not Completed | 10 | 9
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Subject noncompliant | 1 | 3
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment B) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 25 | 24 | 49
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.2 (10.44) | 39.8 (9.37) | 40.5 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Results of Atazanavir (ATV): Treatment A: ATV/Low-Dose Ritonavir (Rtv) 300/100 mg (Results for C0h, Cmin, and Cmax)
Description: The table below shows pharmacokinetic (PK) results of atazanavir (ATZ) when administered as ATV/rtv 300/100 mg pretreatment (Reference) and at Week 2 after treatment (Test). Results are expressed as the predose plasma concentration (C0h), minimum plasma concentration (Cmin), and maximum plasma concentration (Cmax).
Time Frame: Day -1 (Pretreatment); Week 2 (Test)
Population: The population analyzed included all randomized participants with at least 1 etravirine (ETR) intake regardless of their compliance with the protocol (ie, the efficacy ITT population) for which data was available for the PK parameter reported.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- ATV/Rtv 300/100 mg (Reference): Treatment-experienced human immunodeficiency virus - type 1 (HIV-1) infected participants took by mouth atazanavir (ATV)/low-dose ritonavir (rtv) 300/100 mg once daily + 2 nucleoside reverse transcriptase inhibitors (NRTIs) for 14 days during the pre-treatment period. Pharmacokinetic results for ATV provided in the table below are at Day -1.
- ATV/Rtv 300/100 mg (Test): Treatment-experienced human immunodeficiency virus - type 1 (HIV-1) infected participants took by mouth atazanavir (ATV)/low-dose ritonavir (rtv) 300/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 nucleoside reverse transcriptase inhibitor (NRTI) for 48 weeks during the treatment period (Day 1 to Week 48). Pharmacokinetic results for ATV provided in the table below are at Week 2.
Arm/Group | ATV/Rtv 300/100 mg (Reference) | ATV/Rtv 300/100 mg (Test)
Number analyzed (Participants) | 21 | 19
ng/ml
  C0h, ng/ml (Reference, n=21; Test, n=19) | 1339 (1728) | 845.7 (703.3)
  Cmin, ng/ml (Reference, n=20; Test, n=18) | 1104 (1511) | 758.6 (610.5)
  Cmax, ng/ml (Reference, n=20; Test, n=19) | 5652 (2735) | 5232 (2166)
Statistical Analysis 1: Comparison: ATV/Rtv 300/100 mg (Reference) vs ATV/Rtv 300/100 mg (Test); Parameter: minimum plasma concentration (Cmin); Test type: Superiority or Other; Linear mixed effects model; A linear mixed effects model was used controlling for treatment as fixed effect, and participant as a random effect; Least Squares (LS) Means Ratio = 0.82, 90% CI 2-sided [0.55 to 1.22]
Statistical Analysis 2: Comparison: ATV/Rtv 300/100 mg (Reference) vs ATV/Rtv 300/100 mg (Test); Parameter: maximum plasma concentration (Cmax); Test type: Superiority or Other; Linear mixed effects model; A linear mixed effects model was used controlling for treatment as fixed effect, and participant as a random effect; Least Squares (LS) Mean Ratio = 0.96, 90% CI 2-sided [0.80 to 1.16]

2. Primary Outcome: Pharmacokinetic Results of Atazanavir (ATV): Treatment A: ATV/Low-Dose Ritonavir (Rtv) 300/100 mg (Results for AUC24hr)
Description: The table below shows pharmacokinetic (PK) results of atazanavir (ATZ) when administered as ATV/rtv 300/100 mg pretreatment (Reference) and at Week 2 after treatment (Test). Results are expressed as the area under the plasma concentration-time curve from time of intake to 24 hours after dosing (AUC24hr).
Time Frame: Day -1 (Pretreatment); Week 2 (Test)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | ATV/Rtv 300/100 mg (Reference) | ATV/Rtv 300/100 mg (Test)
Number analyzed (Participants) | 19 | 18
ng.h/mL | 60030 (39690) | 55070 (21860)
Statistical Analysis 1: Comparison: ATV/Rtv 300/100 mg (Reference) vs ATV/Rtv 300/100 mg (Test); Parameter: area under the plasma concentration-time curve from time of intake to 24 hours after dosing (AUC24hr); Test type: Superiority or Other; Linear mixed effects model; linear mixed effects model was used controlling for treatment as fixed effect, and participant as a random effect; Least Squares (LS) Means Ratio = 0.96, 90% CI 2-sided [0.76 to 1.22]

3. Primary Outcome: Pharmacokinetic Results of Atazanavir (ATV): Treatment B: ATV/Low-Dose Ritonavir (Rtv) 400/100 mg (Results for C0h, Cmin, and Cmax)
Description: The table below shows pharmacokinetic (PK) results of atazanavir (ATV) when administered as ATV/ritonavir (rtv) 300/100 mg pretreatment (Reference) and when administered as ATV/rtv 400/100 mg at Week 2 after treatment (Test). Results are expressed as the predose plasma concentration (C0h), minimum plasma concentration (Cmin), maximum plasma concentration (Cmax), and area under the plasma concentration-time curve from time of intake to 24 hours after dosing (AUC24hr).
Time Frame: Day -1 (Reference); Week 2 (Test)
Population: The population analyzed included all randomized participants with at least 1 etravirine (ETR) intake regardless of their compliance with the protocol (ie, the efficacy ITT population).
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- ATV/Rtv 400/100 mg (Test): Treatment-experienced human immunodeficiency virus - type 1 (HIV-1) infected participants took by mouth atazanavir (ATV)/ritonavir (rtv) 400/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 nucleoside reverse transcriptase inhibitor (NRTI) for 48 weeks (Day 1 to Week 48). Pharmacokinetic results for ATV provided in the table below are at Week 2.
Arm/Group | ATV/Rtv 300/100 mg (Reference) | ATV/Rtv 400/100 mg (Test)
Number analyzed (Participants) | 21 | 20
ng/ml
  C0h, ng/ml (Reference, n=22; Test, n=20) | 1898 (2298) | 1545 (1296)
  Cmin, ng/ml (Reference, n=21;Test, n=18) | 1671 (2310) | 1107 (866.8)
  Cmax, ng/ml (Reference, n=22; Test, n=20) | 6419 (2853) | 6950 (2693)
Statistical Analysis 1: Comparison: ATV/Rtv 300/100 mg (Reference) vs ATV/Rtv 400/100 mg (Test); Parameter: Minimum plasma concentration (Cmin); Test type: Superiority or Other; Linear mixed effects model; A linear mixed effects model was used controlling for treatment as fixed effect, and participant as a random effect; Least Squares (LS) Means Ratio = 0.91, 90% CI 2-sided [0.63 to 1.33]
Statistical Analysis 2: Comparison: ATV/Rtv 300/100 mg (Reference) vs ATV/Rtv 400/100 mg (Test); Parameter: maximum plasma concentration (Cmax); Test type: Superiority or Other; Linear mixed effects model; A linear mixed effects model was used controlling for treatment as fixed effect, and participant as a random effect; Least Squares (LS) Means Ratio = 1.05, 90% CI 2-sided [0.86 to 1.27]

4. Primary Outcome: Pharmacokinetic Results of Atazanavir (ATV): Treatment B: ATV/Low-Dose Ritonavir (Rtv) 400/100 mg (Results for AUC24hr)
Description: The table below shows pharmacokinetic (PK) results of atazanavir (ATV) when administered as ATV/ritonavir (rtv) 300/100 mg pretreatment (Reference) and when administered as ATV/rtv 400/100 mg at Week 2 after treatment (Test). Results are expressed as the area under the plasma concentration-time curve from time of intake to 24 hours after dosing (AUC24hr).
Time Frame: Day -1 (Reference); Week 2 (Test)
Population: The population analyzed included all randomized participants with at least 1 etravirine (ETR) intake regardless of their compliance with the protocol (ie, the efficacy ITT population) for which data was available for the parameter reported.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | ATV/Rtv 300/100 mg (Reference) | ATV/Rtv 300/100 mg (Test)
Number analyzed (Participants) | 21 | 19
ng.h/mL | 74210 (55480) | 72220 (34600)
Statistical Analysis 1: Comparison: ATV/Rtv 300/100 mg (Reference) vs ATV/Rtv 300/100 mg (Test); Parameter: area under the plasma concentration-time curve from time of intake to 24 hours after dosing (AUC24hr); Test type: Superiority or Other; Llinear mixed effects model; A linear mixed effects model was used controlling for treatment as fixed effect, and participant as a random effect; Least Squares (LS) Means Ratio = 0.99, 90% CI 2-sided [0.81 to 1.21]

5. Primary Outcome: Pharmacokinetic Results of Low-Dose Ritonavir (Rtv): Treatment A: Atazanavir (ATV)/Rtv 300/100 mg (Results for C0h, Cmin, and Cmax)
Description: The table below shows the pharmacokinetic (PK) results of low-dose ritonavir (rtv) when administered as atazanavir (ATV)/rtv 300/100 mg pretreatment (Reference) and at Week 2 after treatment (Test). Results are expressed as the predose plasma concentration (C0h), minimum plasma concentration (Cmin), and maximum plasma concentration (Cmax).
Time Frame: Day -1 (Reference); Week 2 (Test)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | ATV/Rtv 300/100 mg (Reference) | ATV/Rtv 300/100 mg (Test)
Number analyzed (Participants) | 21 | 19
ng/ml
  C0h, ng/ml (Reference, n=21; Test, n=19) | 143.4 (269.8) | 102.5 (157.2)
  Cmin, ng/ml (Reference, n=20; Test, n=18) | 60.42 (73.17) | 43.97 (36.29)
  Cmax, ng/ml (Reference, n=20; Test, n=19) | 1834 (1009) | 1740 (1149)

6. Primary Outcome: Pharmacokinetic Results of Low-Dose Ritonavir (Rtv): Treatment A: Atazanavir (ATV)/Rtv 300/100 mg (Results for AUC24hr)
Description: The table below shows the pharmacokinetic (PK) results of low-dose ritonavir (rtv) when administered as atazanavir (ATV)/rtv 300/100 mg pretreatment (Reference) and at Week 2 after treatment (Test). Results are expressed as the area under the plasma concentration-time curve from time of intake to 24 hours after dosing (AUC24hr).
Time Frame: Day -1 (Reference); Week 2 (Test)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | ATV/Rtv 300/100 mg (Reference) | ATV/Rtv 300/100 mg (Test)
Number analyzed (Participants) | 19 | 18
ng.h/ml | 12560 (6643) | 11120 (6658)

7. Primary Outcome: Pharmacokinetic Results of Low-Dose Ritonavir (Rtv): Treatment B: Atazanavir (ATV)/Rtv 400/100 mg (Results for C0h, Cmin, and Cmax)
Description: The table below shows pharmacokinetic (PK) results of low-dose ritonavir (rtv) when administered as atazanavir (ATV)/ritonavir (rtv) 300/100 mg pretreatment (Reference) and when administered as ATV/rtv 400/100 mg at Week 2 after treatment (Test). Results are expressed as the predose plasma concentration (C0h), minimum plasma concentration (Cmin), maximum plasma concentration (Cmax), and area under the plasma concentration-time curve from time of intake to 24 hours after dosing (AUC24hr).
Time Frame: Day -1 (Reference); Week 2 (Test)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- ATV/Rtv 400/100 mg (Test): Treatment-experienced human immunodeficiency virus - type 1 (HIV-1) infected participants took by mouth atazanavir (ATV)/ritonavir (rtv) 400/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 nucleoside reverse transcriptase inhibitor (NRTI) for 48 weeks (Day 1 to Week 48). Pharmacokinetic results for rtv provided in the table below are at Week 2.
Arm/Group | ATV/Rtv 300/100 mg (Reference) | ATV/Rtv 400/100 mg (Test)
Number analyzed (Participants) | 20 | 19
ng/ml
  C0h, ng/ml (Reference, n=22; Test, n=20) | 109.2 (94.50) | 163.4 (240.2)
  Cmin, ng/ml | 64.70 (51.80) | 75.68 (69.98)
  Cmax, ng/ml (Reference, n=22) | 1882 (1026) | 1847 (859.9)

8. Primary Outcome: Pharmacokinetic Results of Low-Dose Ritonavir (Rtv): Treatment B: Atazanavir (ATV)/Rtv 400/100 mg (Results for AUC24hr)
Description: The table below shows pharmacokinetic (PK) results of low-dose ritonavir (rtv) when administered as atazanavir (ATV)/ritonavir (rtv) 300/100 mg pretreatment (Reference) and when administered as ATV/rtv 400/100 mg at Week 2 after treatment (Test). Results are expressed as the area under the plasma concentration-time curve from time of intake to 24 hours after dosing (AUC24hr).
Time Frame: Day -1 (Reference); Week 2 (Test)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | ATV/Rtv 300/100 mg (Reference) | ATV/Rtv 300/100 mg (Test)
Number analyzed (Participants) | 20 | 19
ng.h/ml | 13880 (8198) | 13660 (6778)

9. Primary Outcome: Pharmacokinetic Results of Etravirine (ETR) (Results for C0h, Cmin, and Cmax)
Description: The table below shows pharmacokinetic (PK) results of ETR in the current study expressed as the predose plasma concentration (C0h), minimum plasma concentration (Cmin) and maximum plasma concentration (Cmax).
Time Frame: Week 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- ATV/Rtv 300/100 mg (Treatment A): Treatment-experienced human immunodeficiency virus - type 1 (HIV-1) infected participants took by mouth atazanavir (ATV)/ritonavir (rtv) 300/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 nucleoside reverse transcriptase inhibitor (NRTI).
- ATV/Rtv 400/100 mg (Treatment B): Treatment-experienced human immunodeficiency virus - type 1 (HIV-1) infected participants took by mouth atazanavir (ATV)/ritonavir (rtv) 400/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 nucleoside reverse transcriptase inhibitor (NRTI).
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment B)
Number analyzed (Participants) | 19 | 20
ng/ml
  C0h (Treatment B, n=19) | 422.2 (327.9) | 316.6 (215.4)
  Cmin (Treatment A, n=16; Treatment B, n=18) | 425.1 (328.1) | 286.5 (198.0)
  Cmax (Treatment A, n=18; Treatment B, n=18) | 773.0 (360.5) | 628.7 (294.0)

10. Primary Outcome: Pharmacokinetic Results of Etravirine (ETR) (Results for AUC12hr)
Description: The table below shows pharmacokinetic (PK) results of ETR in the current study expressed as the area under the plasma concentration-time curve from time of intake to 12 hours after dosing (AUC12hr).
Time Frame: Week 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment B)
Number analyzed (Participants) | 18 | 18
ng.h/mL | 7629 (4213) | 5171 (2695)

11. Primary Outcome: Percentage of Participants With Undetectable Plasma Viral Load (VL) Values (<50 Copies/mL) at Week 48
Description: The table below shows the percentage of participants wih undetectable plasma viral load (VL) values (<50 copies/mL) at Week 48 using the Non-Completing = Failure (NC=F) imputation method (ie, participants who discontinued early were counted as nonresponders by having their VL values after discontinuation imputed with their baseline value, thus resulting in a 0 change).
Time Frame: Week 48
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- ATV/Rtv 300/100 mg (Treatment A): Treatment-experienced human immunodeficiency virus - type 1 (HIV-1) infected participants took by mouth atazanavir (ATV)/ritonavir (rtv) 300/100 mg once daily + 2 nucleoside reverse transcriptase inhibitors (NRTIs) for 2 weeks (Pre-treatment Period) followed by ATV/rtv 300/100 mg once daily + etravine (ETR) 200 mg twice daily + 1 NRTI for 48 weeks (Treatment A).
- ATV/Rtv 400/100 mg (Treatment B): Treatment-experienced human immunodeficiency virus - type 1 (HIV-1) infected participants took by mouth atazanavir (ATV)/ritonavir (rtv) 300/100 mg once daily + 2 nucleoside reverse transcriptase inhibitors (NRTIs) for 2 weeks (Pre-treatment Period) followed by ATV/rtv 400/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 NRTI for 48 weeks (Treatment B).
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment B)
Number analyzed (Participants) | 22 | 22
Percentage of Participants | 50.0 [28.2 to 71.8] | 45.5 [45.5 to 67.8]

12. Secondary Outcome: Change From Prebaseline in CD4+ Cell Count Over Time
Description: The table below shows the mean change from prebaseline over time in CD4+ cell count using the Non-Completing = Failure (NC=F) imputation method.
Time Frame: Prebaseline, Baseline, Weeks 4, 12, 24, 48
Population: as for outcome 3
Measure: Mean (Standard Error); unit: CD4+ cell count
Groups:
- ATV/Rtv 300/100 mg (Treatment A): Treatment-experienced HIV-1 infected participants took by mouth atazanavir (ATV)/low-dose ritonavir (rtv) 300/100 mg once daily + 2 nucleoside reverse transcriptase inhibitors (NRTIs) for 2 weeks (Pre-treatment Period) followed by ATV/rtv 300/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 NRTI for 48 weeks (Treatment A).
- ATV/Rtv 400/100 mg (Treatment B): Treatment-experienced HIV-1 infected participants took by mouth atazanavir (ATV)/low-dose ritonavir (rtv) 300/100 mg once daily + 2 nucleoside reverse transcriptase inhibitors (NRTIs) for 2 weeks (Pre-treatment Period) followed by ATV/rtv 400/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 NRTI for 48 weeks (Treatment B).
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment B)
Number analyzed (Participants) | 22 | 22
CD4+ cell count
  Baseline | 16 (11.8) | 8 (18)
  Week 4 | 55 (15.4) | 46 (27.4)
  Week 12 | 31 (15.0) | 72 (23.5)
  Week 24 | 54 (22.0) | 83 (23.2)
  Week 48 | 105 (31.1) | 132 (32.6)

13. Secondary Outcome: The Percentage of Participants With a Virologic Response Using the Non-Completing = Failure (NC=F) Imputation Method
Description: The table below shows the percentage of participants per time point with a virologic response defined as having a plasma viral load (VL) <50 copies/mL, and with plasma VL <400 copies/mL using the Non-Completing = Failure (NC=F) imputation method (ie, participants who discontinued early were counted as nonresponders by having their VL values after discontinuation imputed with their Baseline value, thus resulting in a 0 change).
Time Frame: Baseline, Weeks 4, 12, 24, 48
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment B)
Number analyzed (Participants) | 22 | 22
Percentage of Participants
  <50 copies/mL, Baseline | 9.1 | 9.1
  <50 copies/mL, Week 4 | 31.8 | 36.4
  <50 copies/mL, Week 12 | 59.1 | 59.1
  <50 copies/mL, Week 24 | 63.6 | 63.6
  <50 copies/mL, Week 48 | 50.0 | 45.5
  <400 copies/mL, Baseline | 40.9 | 40.9
  <400 copies/mL, Week 4 | 77.3 | 77.3
  <400 copies/mL, Week 12 | 68.2 | 81.8
  <400 copies/mL, Week 24 | 72.7 | 72.7
  <400 copies/mL, Week 48 | 50.0 | 59.1

14. Secondary Outcome: The Percentage of Participants With a Virologic Response Using the Time to Loss of Virologic Response (TLOVR) Imputation Method
Description: The table below shows the percentage of participants with a virologic response defined as a viral load <50 Copies/mL and <400 Copies/mL per time point calculated using the time to loss of virologic response (TLOVR) imputation method.
Time Frame: Baseline, Weeks 4, 12, 24, 48
Population: as for outcome 3
Measure: Number; unit: Percentage of Particpants
Groups:
- ATV/Rtv 400/100 mg (Treatment A): Treatment-experienced HIV-1 infected participants took by mouth atazanavir (ATV)/low-dose ritonavir (rtv) 300/100 mg once daily + 2 nucleoside reverse transcriptase inhibitors (NRTIs) for 2 weeks (Pre-treatment Period) followed by ATV/rtv 400/100 mg once daily + etravirine (ETR) 200 mg twice daily + 1 NRTI for 48 weeks (Treatment B).
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment A)
Number analyzed (Participants) | 22 | 22
Percentage of Particpants
  <50 copies/mL, Baseline | 9.1 | 4.5
  <50 copies/mL, Week 4 | 31.8 | 36.4
  <50 copies/mL, Week 12 | 59.1 | 54.5
  <50 copies/mL, Week 24 | 63.6 | 59.1
  <50 copies/mL, Week 48 | 45.5 | 50.0
  <400 copies/mL, Baseline | 36.4 | 40.9
  <400 copies/mL, Week 4 | 77.3 | 77.3
  <400 copies/mL, Week 12 | 68.2 | 86.4
  <400 copies/mL, Week 24 | 68.2 | 68.2
  <400 copies/mL, Week 48 | 59.1 | 54.5

15. Secondary Outcome: The Percentage of Participants With a Virologic Response (Plasma Viral Load < 50 Copies/mL) at Week 48 Using the Snapshot Analysis Method
Description: The table below provides the results from the snapshot analysis method that includes the percentage of participants with virologic response (<50 copies/mL), the percentage of participants who were virologic failures (VF) (>50 copies/mL, discontinued prior to time X for reasons of VF or for other reasons, except for VF or adverse event, with a last viral load >50 copies/mL), and the percentage of participants with no viral load (VL) data available at Week 48.
Time Frame: Week 48
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment B)
Number analyzed (Participants) | 22 | 22
Percentage of Participants
  Virologic Response | 50.0 | 45.5
  Virologic Failure | 31.8 | 36.4
  No VL Data Available | 18.2 | 18.2

16. Secondary Outcome: Change From Pre-Baseline in Log10 Viral Load Over Time
Description: The table below shows the mean change from prebaseline over time in log10 (Copies/mL) plasma viral load using the Non-Completing = Failure (NC=F) imputation method.
Time Frame: Pre-Baseline, Baseline, Weeks 4, 12, 24, 48
Population: as for outcome 3
Measure: Mean (Standard Error); unit: log10 (Copies/mL)
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment B)
Number analyzed (Participants) | 22 | 22
log10 (Copies/mL)
  Baseline | -1.4 (0.14) | -1.4 (0.18)
  Week 4 | -1.9 (0.18) | -1.8 (0.15)
  Week 12 | -1.7 (0.26) | -2.0 (0.23)
  Week 24 | -1.8 (0.24) | -1.8 (0.27)
  Week 48 | -1.4 (0.24) | -1.4 (0.29)

17. Secondary Outcome: Time to Confirmed Virologic Response
Description: The table below provides the time in days it took participants to reach a confirmed virologic response defined as a plasma viral load (VL) <50 copies/mL, and plasma VL <400 copies/mL analyzed according to the Time to Loss of Virologic Response (TLOVR) imputation method.
Time Frame: Prebaseline to Week 48
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment B)
Number analyzed (Participants) | 22 | 22
Days
  Plasma VL < 50 copies/mL | 71.0 (10.87) [44.0 to 129.0] | 76.0 (9.95) [42.0 to 99.0]
  Plasma VL < 400 copies/mL | 28.0 (5.02) [15.0 to 43.0] | 28.0 (6.47) [15.0 to 43.0]

18. Secondary Outcome: Time to Virologic Failure
Description: The table below shows the number of days to virologic failure defined as a plasma viral load (VL) > 50 copies/mL for participants who had been virologic responders (ie, having a plasma VL <50, and <400 copies/mL according to the time to loss of virologic response [TLOVR] imputation method). Time to virologic failure was the time to subsequent loss of virologic response, and the time was calculated from Prebaseline (Week -2). Participants who never achieved a virologic response were defined as nonresponders and counted as virologic failures on Day 1.
Time Frame: Prebaseline to Week 48
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment B)
Number analyzed (Participants) | 22 | 22
Days
  Virologic Responders (Plasma VL < 50 copies/mL) | 318.0 (31.90) [78.0 to NA] — The upper limit of the 95% CI could not be assessed because a sufficient number of participants did not experience virologic failure. | NA (22.46) [NA to NA] — Median cannot be assessed since less than 50% of participants experienced virologic failure.
  Virologic Responders (Plasma VL < 400 copies/mL) | NA (28.92) [NA to NA] — Median cannot be assessed since less than 50% of participants experienced virologic failure | NA (17.28) [NA to NA] — Median cannot be assessed since less than 50% of participants experienced virologic failure

ADVERSE EVENTS:
Time Frame: Up to a maximum of 56 weeks.
Description: To also include the safety data of 6 participants who discontinued during the Pretreatment Period, the safety analyses were performed on the ITT population defined as all participants who had at least 1 atazanavir (ATV)/low dose ritonavir (rtv) intake regardless of their compliance with the protocol (ie, the 'safety ITT population').
Arm/Group | ATV/Rtv 300/100 mg (Treatment A) | ATV/Rtv 400/100 mg (Treatment B)
Serious Adverse Events (participants affected / at risk) | 4/25 | 2/25
Other Adverse Events (participants affected / at risk) | 21/25 | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATV/Rtv 300/100 mg (Treatment A) (N=25) | ATV/Rtv 400/100 mg (Treatment B) (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATV/Rtv 300/100 mg (Treatment A) (N=25) | ATV/Rtv 400/100 mg (Treatment B) (N=25)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 0
Bronchitis (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 2 | 3
Sinusitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Blood bilirubin increased (Investigations) | 3 | 2
Headache (Nervous system disorders) | 3 | 3
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 2 | 2
Anxiety disorder (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is the policy of the sponsor not to allow investigators to publish their results or findings from the study prior to the sponsor's publication of the overall trial results. The investigator agrees that before he/she publishes any results of this trial, he/she shall allow at least 45 days for the sponsor to review the prepublication manuscript prior to submission of the manuscript to the publisher.